CLINICAL TRIAL: NCT05184088
Title: An Open-label, Multi-center, Non-randomized Pivotal Phase 3 Study to Evaluate the Efficacy and Safety of [18F]Florbetaben Positron Emission Tomography (PET) Imaging to Diagnose Cardiac AL Amyloidosis
Brief Title: Efficacy of [18F]Florbetaben PET for Diagnosis of Cardiac AL Amyloidosis
Acronym: CArdiag
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Life Molecular Imaging GmbH (Industry)
Collaborators: pharmtrace klinische Entwicklung GmbH (Unknown)
Responsible Party: Sponsor
Organization: Life Molecular Imaging SA (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FBB-02-01-21
Record Dates: First submitted 2022-01-06; First posted 2022-01-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Amyloidosis; AL Amyloidosis; ATTR Amyloidosis
Keywords: AL Amyloidosis; ATTR Amyloidosis; Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Immunoglobulin Light-chain Amyloidosis | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Intervention Model Description: All eligible patients will receive a single administration of the imaging agent [18F]florbetaben at a radioactive dose of 300 MBq.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with suspected cardiac amyloidosis (Experimental): After enrolment, patients will be subjected to diagnostic procedures according to standard of care to resolve diagnostic uncertainties and to clarify possible cardiac involvement. The results of the clinical work-up will be used a standard of truth, i.e. patients with initially suspected cardiac amyloidosis that where subsequently clinically diagnosed with cardiac AL Amyloidosis, cardiac ATTR Amyloidosis, other cardiac Amyloidosis or non cardiac amyloidosis.
  Interventions: Drug: [18F]florbetaben

INTERVENTIONS:
Drug: [18F]florbetaben — All enrolled patients will undergo [18F]florbetaben PET imaging.
  Other Names: Neuraceq

SUMMARY:
This is an open-label, multi-center pivotal Phase 3 study to visually and quantitatively assess PET images obtained after single application of 300 MBq [18F]florbetaben and PET scanning of patients with suspected cardiac amyloidosis.

DETAILED DESCRIPTION:
This is an open-label, multi-center pivotal Phase 3 study to visually and quantitatively assess PET images obtained after single application of 300 MBq [18F]florbetaben and PET scanning of patients with suspected cardiac amyloidosis or with a putative diagnosis of cardiac amyloidosis but with remaining diagnostic uncertainty (e.g., unclear etiology or cardiac manifestation) or patients with diagnosis of amyloidosis but unclear cardiac involvement.

The diagnostic efficacy of the visual and quantitative assessments of [18F]florbetaben PET images for diagnosis of cardiac AL Amyloidosis will be determined by comparison to the standard of truth (SoT) obtained through standard of care clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age ≥18 years
* Able to understand, sign and date written informed consent
* Written informed consent must be obtained before any study procedures are performed
* Subjects being considered for a possible diagnosis of cardiac amyloidosis by
* 1. One of the following conditions:

  * Established systemic amyloidosis without proven cardiac involvement,
  * Known plasma cell dyscrasia (MGUS, multiple myeloma),
  * Pathological free light chain levels in urine or serum,
  * Presence of heart failure with preserved ejection fraction
* 2. AND one of the following parameters, indicative of cardiac manifestation:

  * Mean (left ventricular (LV) wall + septum) thickness >12mm as measured by echocardiography or CMR in absence of other known cause of left ventricular hypertrophy (LVH),
  * NT-proBNP >335 ng/L (in case a value for NT-proBNP is not available, BNP > 81ng/L may be used instead)
* Planned diagnostic procedure to establish diagnosis and cardiac involvement (e.g., endomyocardial biopsy or extracardiac biopsy in conjunction with cardiac magnetic resonance imaging/echocardiography or bone scintigraphy)
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or post-menopausal for at least 1 year (no menses for 12 months without an alternative medical cause). If they are of child-bearing potential, they must commit to use of a highly effective contraceptive measure for at least one week following the PET scan (including combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilaterial tubal occlusion, vasectomised parner or secual abstinence).
* Male subjects and their partners of childbearing potential must commit to the use of a highly effective method of contraception for a minimum of 90 days following the PET scan (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilaterial tubal occlusion, male subjects with vasectomy or sexual abstinence)
* Male subjects must commit to not donate sperm for a minimum of 90 days after the PET scan

Exclusion Criteria:

* Any known allergic reactions or hypersensitivity towards any compound of the study drug
* Severe hepatic impairment (AST/ALT >5 x ULN; bilirubin >3 x ULN)
* Inability to lay flat for up to 60 min
* Pregnant, lactating or breastfeeding
* Unwilling and/or unable to cooperate with study procedures
* Having been administered a radiopharmaceutical within 10 radioactive half-lives prior to study drug administration in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the visual assessment of [18F]florbetaben PET images for the diagnosis of cardiac AL amyloidosis. | Up to 12 weeks
  The results from the visual assessment of [18F]florbetaben PET images are compared to the clinical diagnosis established through histological verification of the presence or absence of AL amyloidosis with cardiac involvement determined either through endomyocardial biopsy or through extracardiac biopsy in conjunction with typical CMR or echocardiography imaging features as the standard of truth.

SECONDARY OUTCOMES:
Sensitivity and specificity of [18F]florbetaben PET for the diagnosis of cardiac AL amyloidosis using quantification. | Up to 12 weeks
  The sensitivity and specificity of [18F]florbetaben PET for the diagnosis of cardiac AL amyloidosis will be determined by using quantitative image analysis.
Correlation of quantitative [18F]florbetaben PET results with left ventricular ejection fraction (LV EF) and left ventricular mass (LV mass). | Up to 12 weeks
  Correlation of quantitative [18F]florbetaben PET results with left ventricular ejection fraction (LV EF) and left ventricular mass (LV mass).
Correlation of quantitative [18F]florbetaben PET results with AL CA stage I - IV based on FLC-diff, cTnT and NT-proBNP levels. | Up to 12 weeks
  Correlation of quantitative [18F]florbetaben PET results with AL CA stage I - IV based on FLC-diff, cTnT and NT-proBNP levels.
Impact of PET imaging (AL-CA/non AL-CA) on diagnostic thinking and patient management will be assessed with physician's questionnaires before and after the diagnostic work-up, and after receipt of the PET results. | Up to 14 weeks
  The impact of PET imaging (AL-CA/non AL-CA) on diagnostic thinking and patient management will be assessed with physician's questionnaires before and after the diagnostic work-up, and after receipt of the PET results.
Number of adverse events | Up to 17 days after imaging visit
  Safety will be evaluated by collection of Adverse Events.

OTHER OUTCOMES:
Sensitivity and specificity of [18F]florbetaben PET images for a differential diagnosis between AL CA, ATTR CA and non CA will be assessed. | Up to 12 weeks
  In this exploratory endpoint the sensitivity and specificity of [18F]florbetaben PET images for a differential diagnosis between AL CA, ATTR CA and non CA will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Stephens, MD, PhD, Study Director — Life Molecular Imaging
Locations (14):
- United States (3):
  - St Luke's Hospital, Kansas City, Kansas
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Germany (6):
  - University of Augsburg, Augsburg
  - Charite Berlin, Berlin
  - University of Essen, Essen
  - HOPA Hamburg, Hamburg
  - University of Heidelberg, Heidelberg
  - University of Würzburg, Würzburg
- Spain (4):
  - Hospital University Bellvitge, Barcelona
  - Hospital University Puerta de Hierro, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - University of Salamanca, Salamanca
- Royal Free Hospital, London, United Kingdom